CLINICAL TRIAL: NCT05239221
Title: A Single and Multiple Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AZP-3601, a Synthetic Parathyroid Hormone Analog, in Healthy Subjects and in Subjects With Hypoparathyroidism
Brief Title: AZP-3601 SAD and MAD Study in Healthy Subjects and Patients With Hypoparathyroidism
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Amolyt Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AZP-3601-CLI-001
Record Dates: First submitted 2022-01-07; First posted 2022-02-14 (Actual); Results first posted 2024-01-31 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Chronic Hypoparathyroidism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part C is open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AZP-3601 (Experimental): subcutaneous (sc) administration once daily
  Interventions: Drug: AZP-3601
- Placebo (Parts A and B) (Placebo Comparator): subcutaneous (sc) administration once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZP-3601 — Lyophilized powder of AZP-3601 to be reconstituted with water for injection before injection
  Other Names: eneboparatide
  Arms: AZP-3601
Drug: Placebo — Saline solution visually matching active medication
  Arms: Placebo (Parts A and B)

SUMMARY:
This study is investigating the safety, tolerability, pharmacodynamics and pharmacokinetics of AZP-3601 following single and repeated administration in both healthy volunteers and patients with chronic hypoparathyroidism (cHP)

The protocol includes 3 parts:

* Part A: first-in-human single ascending dose (SAD) study in healthy volunteers
* Part B: multiple ascending dose (MAD) study with 2 weeks of treatment in healthy volunteers
* Part C: open-label MAD study with a total treatment duration of 3 months in patients with cHP.

ELIGIBILITY:
Main inclusion criteria

* Part A: healthy male volunteers aged 18 to 60 years old inclusive with a body mass index of 19 to 28 kg/m2
* Part B: healthy male and female volunteers (non-child bearing potential) aged 18 to 60 years inclusive with a Body mass index of 19 to 28 kg/m2
* Part C:

  1. Male and female patients aged 18 to 75 years inclusive
  2. History of cHP for ≥12 months at the time of screening with documentation of two measurements of serum calcium and parathyroid hormone (PTH).
  3. Requirement for therapy with calcitriol ≥0.25 μg per day or alphacalcidol ≥0.50 μg per day (both are active vitamin D supplements), and requirement for supplemental oral calcium treatment ≥1000 mg per day over and above normal dietary calcium intake at baseline assessments.

Main exclusion criteria

* Parts A and B:

  1. Clinically significant abnormal lab values, as judged by the investigator
  2. Using tobacco products with 3 months prior to first drug administration
  3. History of alcohol abuse or drug addiction
* Part C:

  1. Known history of autosomal-dominant hypocalcemia (ADH resulting from gain-of-function calcium-sensing receptor [CaSR] or GNA11 mutations) or pseudohypoparathyroidism (impaired responsiveness to PTH)
  2. Any current disease that might affect calcium metabolism or calcium phosphate homeostasis other than HP
  3. Use of medications such as loop and thiazide diuretics, raloxifene hydrochloride, lithium, methotrexate, cardiac glycosides (e.g., digoxin or digitoxin) or systemic corticosteroids within 4 weeks prior to start of treatment.
  4. Previous treatment with PTH-like drugs, including PTH(1-84), PTH(1-34), or abaloparatide, within 3 months prior to screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Amolyt Pharma Investigational Site Hungary, Budapest, Hungary
- PRA-EDS, Groningen, Netherlands

REFERENCES:
- [Derived] Ovize M, Allas S, Culler MD, Milano S, Ouldrouis T, Sumeray M, van de Wetering de Rooij J, Mannstadt M. Phase 1 clinical trial of eneboparatide, a novel PTH receptor 1 agonist. Endocr Connect. 2025 Jun 19;14(6):e240464. doi: 10.1530/EC-24-0464. Print 2025 Jun 1. PMID 40423237

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 132 subjects were enrolled in the study. Of those, 52 subjects were enrolled in Part A (Phase 1), 52 subjects were enrolled in Part B (Phase 1), and 28 subjects were enrolled in Part C (Phase 2a).
Groups:
- Part A (Cohort A1, 5 ug Dose): Healthy volunteers were administered a single subcutaneous (SC) dose of 5ug of AZP-3601 on Day 1.
- Part A (Cohort A2, 10 ug Dose): Healthy volunteers were administered a single subcutaneous (SC) dose of 10 ug of AZP-3601 on Day 1.
- Part A (Cohort A3, 20 ug Dose): Healthy volunteers were administered a single subcutaneous (SC) dose of 20 ug of AZP-3601 on Day 1.
- Part A (Cohort A4, 40 ug Dose): Healthy volunteers were administered a single subcutaneous (SC) dose of 40 ug of AZP-3601 on Day 1.
- Part A (Cohort A5, 60 ug Dose): Healthy volunteers were administered a single subcutaneous (SC) dose of 60 ug of AZP-3601 on Day 1.
- Part A (Cohort A6, 120 ug Dose): Healthy volunteers were administered a single subcutaneous (SC) dose of 120 ug of AZP-3601 on Day 1.
- Part A (Cohort A7, 90 ug Dose): Healthy volunteers were administered a single subcutaneous (SC) dose of 90 ug of AZP-3601 on Day 1.
- Part A (Placebo): Healthy volunteers were administered a single, subcutaneous dose of placebo on Day 1.
- Part B (Cohort B1, 10 ug Doses): Healthy volunteers were administered a multiple subcutaneous (SC) doses of 10 ug of AZP-3601, once daily, from Day 1 to Day 14.
- Part B (Cohort B2, 20 ug Doses): Healthy volunteers were administered a multiple subcutaneous (SC) doses of 20 ug of AZP-3601, once daily, from Day 1 to Day 14.
- Part B (Cohort B3, 40 ug Doses): Healthy volunteers were administered a multiple subcutaneous (SC) doses of 40 ug of AZP-3601, once daily, from Day 1 to Day 14.
- Part B (Cohort B4, 60 ug Doses): Healthy volunteers were administered a multiple subcutaneous (SC) doses of 60 ug of AZP-3601, once daily, from Day 1 to Day 14.
- Part B (Cohort B5, 80 ug Doses): Healthy volunteers were administered a multiple subcutaneous (SC) doses of 80 ug of AZP-3601, once daily, from Day 1 to Day 14.
- Part B (Placebo): Healthy volunteers were administered a multiple subcutaneous (SC) doses of placebo, once daily, from Day 1 to Day 14.
- Part C (Cohort C1, Starting Dose of 20 ug/Day): Patients with hypoparathyroidism were treated with a once daily subcutaneous doses of AZP-3601 from Day 1 to Day 84. The starting dose was 20 ug/day, and up-titration of the dose was allowed from Day 14 onwards.
- Part C (Cohort C2, Starting Dose of 10 ug/Day): Patients with hypoparathyroidism were treated with a once daily subcutaneous doses of AZP-3601 from Day 1 to Day 84. The starting dose was 10 ug/day, and up-titration of the dose was allowed from Day 14 onwards.
Period: Overall Study
Arm/Group | Part A (Cohort A1, 5 ug Dose) | Part A (Cohort A2, 10 ug Dose) | Part A (Cohort A3, 20 ug Dose) | Part A (Cohort A4, 40 ug Dose) | Part A (Cohort A5, 60 ug Dose) | Part A (Cohort A6, 120 ug Dose) | Part A (Cohort A7, 90 ug Dose) | Part A (Placebo) | Part B (Cohort B1, 10 ug Doses) | Part B (Cohort B2, 20 ug Doses) | Part B (Cohort B3, 40 ug Doses) | Part B (Cohort B4, 60 ug Doses) | Part B (Cohort B5, 80 ug Doses) | Part B (Placebo) | Part C (Cohort C1, Starting Dose of 20 ug/Day) | Part C (Cohort C2, Starting Dose of 10 ug/Day)
Started | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 13 | 8 | 8 | 10 | 8 | 8 | 10 | 12 | 16
Completed | 3 | 6 | 6 | 6 | 6 | 6 | 5 | 13 | 8 | 8 | 8 | 7 | 8 | 10 | 12 | 15
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A (Cohort A1, 5 ug Dose) | Part A (Cohort A2, 10 ug Dose) | Part A (Cohort A3, 20 ug Dose) | Part A (Cohort A4, 40 ug Dose) | Part A (Cohort A5, 60 ug Dose) | Part A (Cohort A6, 120 ug Dose) | Part A (Cohort A7, 90 ug Dose) | Part A (Placebo) | Part B (Cohort B1, 10 ug Doses) | Part B (Cohort B2, 20 ug Doses) | Part B (Cohort B3, 40 ug Doses) | Part B (Cohort B4, 60 ug Doses) | Part B (Cohort B5, 80 ug Doses) | Part B (Placebo) | Part C (Cohort C1, Starting Dose of 20 ug/Day) | Part C (Cohort C2, Starting Dose of 10 ug/Day) | Total
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 13 | 8 | 8 | 10 | 8 | 8 | 10 | 12 | 16 | 132
Age, Continuous [Mean (Full Range); unit: years] | 29.3 [28 to 30] | 38.8 [20 to 59] | 23.7 [19 to 33] | 30.0 [20 to 60] | 26.3 [20 to 50] | 21.0 [18 to 24] | 35.3 [23 to 58] | 29.2 [18 to 57] | 38.3 [19 to 59] | 42.9 [28 to 60] | 39.7 [19 to 59] | 30.1 [19 to 43] | 33.3 [20 to 48] | 32.0 [22 to 57] | 62.7 [44 to 72] | 54.0 [26 to 72] | 37.9 [18 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 9 | 12 | 25
  Male | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 13 | 8 | 6 | 9 | 8 | 8 | 9 | 3 | 4 | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 3 | 0 | 0 | 9
  Not Hispanic or Latino | 3 | 6 | 6 | 6 | 6 | 5 | 6 | 12 | 8 | 8 | 9 | 7 | 6 | 7 | 12 | 15 | 122
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 3
  White | 3 | 5 | 5 | 5 | 5 | 5 | 6 | 10 | 8 | 5 | 10 | 7 | 3 | 7 | 12 | 16 | 112
  More than one race | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hungary | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 6 | 15
  Spain | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 7
  France | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
  Netherlands | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 13 | 8 | 8 | 10 | 8 | 8 | 10 | 0 | 0 | 104

OUTCOME MEASURES:

1. Primary Outcome: Treatment Emergent Adverse Events (TEAEs)
Description: Number of Treatment Emergent Adverse Events (TEAEs), as assessed by medDRA (v25).
Time Frame: Up to 2 weeks in Part A and Part B, and up to 3 months in Part C
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Cohort A1, 5 ug Dose) | Part A (Cohort A2, 10 ug Dose) | Part A (Cohort A3, 20 ug Dose) | Part A (Cohort A4, 40 ug Dose) | Part A (Cohort A5, 60 ug Dose) | Part A (Cohort A6, 120 ug Dose) | Part A (Cohort A7, 90 ug Dose) | Part A (Placebo) | Part B (Cohort B1, 10 ug Doses) | Part B (Cohort B2, 20 ug Doses) | Part B (Cohort B3, 40 ug Doses) | Part B (Cohort B4, 60 ug Doses) | Part B (Cohort B5, 80 ug Doses) | Part B (Placebo) | Part C (Cohort C1, Starting Dose of 20 ug/Day) | Part C (Cohort C2, Starting Dose of 10 ug/Day)
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 13 | 8 | 8 | 10 | 8 | 8 | 10 | 12 | 16
Participants | 2 | 3 | 5 | 1 | 3 | 6 | 6 | 8 | 6 | 7 | 10 | 8 | 7 | 9 | 7 | 12

2. Secondary Outcome: Observed Maximum Concentration (Cmax) - Part A
Description: Observed maximum concentration (Cmax) of AZP-3601 (pg/mL) in Part A
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Part A (Cohort A1, 5 ug Dose) | Part A (Cohort A2, 10 ug Dose) | Part A (Cohort A3, 20 ug Dose) | Part A (Cohort A4, 40 ug Dose) | Part A (Cohort A5, 60 ug Dose) | Part A (Cohort A6, 120 ug Dose) | Part A (Cohort A7, 90 ug Dose)
Number analyzed (Participants) | 2 | 4 | 6 | 3 | 6 | 6 | 6
pg/mL | 6.82 (2.19) | 11.4 (4.32) | 24.1 (8.18) | 26.3 (4.79) | 28.5 (10.8) | 57.4 (28.7) | 37.5 (11.6)

3. Secondary Outcome: Observed Maximum Concentration (Cmax) - Part B
Description: Observed maximum concentration (Cmax) of AZP-3601 (pg/mL) in Part B
Time Frame: Day 1, Day 14
Population: Data not collected for a few subjects (missing data or site error)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Part B (Cohort B1, 10 ug Doses) | Part B (Cohort B2, 20 ug Doses) | Part B (Cohort B3, 40 ug Doses) | Part B (Cohort B4, 60 ug Doses) | Part B (Cohort B5, 80 ug Doses)
Number analyzed (Participants) | 4 | 8 | 8 | 8 | 8
pg/mL
  Day 1 | 20.6 (3.43) | 19.6 (5.68) | 23.8 (8.97) | 42.9 (30.3) | 124 (105)
  Day 14: number analyzed (Participants) | 4 | 7 | 8 | 7 | 8
  Day 14 | 18.4 (5.37) | 18.3 (6.78) | 23.6 (5.50) | 44.9 (17.9) | 63.5 (28.3)

4. Secondary Outcome: Observed Maximum Concentration (Cmax) - Part C
Description: Observed maximum concentration (Cmax) of AZP-3601 (pg/mL) in Part C.
Time Frame: Day 1, Day 14, Day 28, Day 84
Population: One (1) subject dropped out in Cohort 2 prior to the extension phase and one (1) subject from Cohort 2 did not participate in the extension phase (data on Day 84). In addition, data not collected for a few subjects (missing data or site error). PK data was not collected in Cohort 1 on Day 84 per the protocol at the time. The protocol was updated following completion of Cohort 1 to collect PK information in Cohort 2 on Day 84.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Part C (Cohort C1, Starting Dose of 20 ug/Day) | Part C (Cohort C2, Starting Dose of 10 ug/Day)
Number analyzed (Participants) | 12 | 16
pg/mL
  Day 1: number analyzed (Participants) | 12 | 15
  Day 1 | 21.3 (9.20) | 11.9 (7.82)
  Day 14: number analyzed (Participants) | 12 | 14
  Day 14 | 22.3 (11.7) | 10.4 (7.73)
  Day 28: number analyzed (Participants) | 12 | 15
  Day 28 | 18.4 (7.42) | 21.5 (17.9)
  Day 84: number analyzed (Participants) | 0 | 10
  Day 84 |  | 89.9 (63.9)

5. Secondary Outcome: Area Under the Plasma-drug Concentration Time Curve (AUC) - Part A
Description: Area under the plasma-drug concentration time curve (AUC) (pg*h/mL) in Part A
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Part A (Cohort A1, 5 ug Dose) | Part A (Cohort A2, 10 ug Dose) | Part A (Cohort A3, 20 ug Dose) | Part A (Cohort A4, 40 ug Dose) | Part A (Cohort A5, 60 ug Dose) | Part A (Cohort A6, 120 ug Dose) | Part A (Cohort A7, 90 ug Dose)
Number analyzed (Participants) | 2 | 4 | 6 | 3 | 6 | 6 | 6
pg*h/mL | 0.399 (0.032) | 5.20 (3.38) | 9.55 (4.12) | 10.4 (13.4) | 16.8 (14.7) | 26.1 (16.4) | 31.7 (12.5)

6. Secondary Outcome: Area Under the Plasma-drug Concentration Time Curve (AUC) - Part B
Description: Area Under the Plasma-drug Concentration Time Curve (AUC) (pg*h/mL) in Part B
Time Frame: Day 1, Day 14
Population: Data not collected for a few subjects (missing data or site error).
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Part B (Cohort B1, 10 ug Doses) | Part B (Cohort B2, 20 ug Doses) | Part B (Cohort B3, 40 ug Doses) | Part B (Cohort B4, 60 ug Doses) | Part B (Cohort B5, 80 ug Doses)
Number analyzed (Participants) | 4 | 8 | 8 | 8 | 8
pg*h/mL
  Day 1 | 3.26 (3.20) | 7.69 (5.52) | 15.8 (11.5) | 43.3 (18.1) | 64.2 (56.1)
  Day 14: number analyzed (Participants) | 4 | 7 | 8 | 7 | 8
  Day 14 | 2.02 (2.41) | 4.63 (3.29) | 12.5 (4.75) | 58.8 (30.3) | 51.9 (51.6)

7. Secondary Outcome: Area Under the Plasma-drug Concentration Time Curve (AUC) - Part C
Description: Area Under the Plasma-drug Concentration Time Curve (AUC) (pg*h/mL) in Part C.
Time Frame: Day 1, Day 14, Day 28, Day 84
Population: One (1) subject dropped out in Cohort 2 prior to the extension phase and one (1) subject from Cohort 2 did not participate in the extension phase (data on Day 84). In addition, data not collected for a few subjects (missing data or site error). Pharmacokinetic (PK) data was not collected in Cohort 1 on Day 84 per the protocol at the time. The protocol was updated following completion of Cohort 1 to collect PK information in Cohort 2 on Day 84.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Part C (Cohort C1, Starting Dose of 20 ug/Day) | Part C (Cohort C2, Starting Dose of 10 ug/Day)
Number analyzed (Participants) | 12 | 16
pg*h/mL
  Day 1: number analyzed (Participants) | 12 | 15
  Day 1 | 11.9 (9.53) | 4.90 (4.87)
  Day 14: number analyzed (Participants) | 12 | 14
  Day 14 | 16.1 (14.0) | 3.99 (4.22)
  Day 28: number analyzed (Participants) | 12 | 15
  Day 28 | 12.7 (7.58) | 11.8 (11.1)
  Day 84: number analyzed (Participants) | 0 | 10
  Day 84 |  | 116 (111)

8. Secondary Outcome: Calcium Corrected for Albumin - Part A
Description: Levels of calcium corrected for albumin (mg/dL) in Part A
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part A (Cohort A1, 5 ug Dose) | Part A (Cohort A2, 10 ug Dose) | Part A (Cohort A3, 20 ug Dose) | Part A (Cohort A4, 40 ug Dose) | Part A (Cohort A5, 60 ug Dose) | Part A (Cohort A6, 120 ug Dose) | Part A (Cohort A7, 90 ug Dose) | Part A (Placebo)
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 13
mg/dL | 9.700 (0.0800) | 9.375 (0.6215) | 9.688 (0.3448) | 9.782 (0.4303) | 10.065 (0.2934) | 10.293 (0.5258) | 10.195 (0.2601) | 9.634 (0.3030)

9. Secondary Outcome: Calcium Corrected for Albumin - Part B
Description: Levels of calcium corrected for albumin (mg/dL) in Part B
Time Frame: 24 hours, Day 14
Population: One (1) subject in Cohort B4 discontinued from the study.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part B (Cohort B1, 10 ug Doses) | Part B (Cohort B2, 20 ug Doses) | Part B (Cohort B3, 40 ug Doses) | Part B (Cohort B4, 60 ug Doses) | Part B (Cohort B5, 80 ug Doses) | Part B (Placebo)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 10
mg/dL
  24 hours | 9.818 (0.3283) | 9.661 (0.3492) | 10.121 (0.4320) | 10.01 (0.30) | 10.01 (0.41) | 9.68 (0.21)
  Day 14: number analyzed (Participants) | 8 | 8 | 8 | 7 | 8 | 10
  Day 14 | 9.586 (0.3173) | 9.650 (0.2081) | 10.055 (0.5916) | 10.06 (0.59) | 10.94 (0.97) | 9.79 (0.24)

10. Secondary Outcome: Calcium Corrected for Albumin - Part C
Description: Levels of calcium corrected for albumin (mg/dL) in Part C.
Time Frame: Day 1, Day 14, Day 28 and Day 84
Population: One (1) subject dropped out in Cohort 2 prior to the extension phase. In addition to this subject, two (2) subjects from Cohort 1 and one (1) subject from Cohort 2 did not participate in the extension phase (data on Day 84). In addition, data not collected for a few subjects (missing data or site error).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part C (Cohort C1, Starting Dose of 20 ug/Day) | Part C (Cohort C2, Starting Dose of 10 ug/Day)
Number analyzed (Participants) | 12 | 16
mg/dL
  Day 1 (hour 0): number analyzed (Participants) | 11 | 16
  Day 1 (hour 0) | 8.44 (0.420) | 8.61 (0.552)
  Day 14 | 8.48 (0.537) | 8.38 (0.726)
  Day 28: number analyzed (Participants) | 12 | 15
  Day 28 | 8.64 (0.491) | 8.537 (0.697)
  Day 84: number analyzed (Participants) | 10 | 13
  Day 84 | 7.95 (0.817) | 8.73 (0.878)

11. Secondary Outcome: Serum Phosphate - Part A
Description: Serum phosphate levels (mg/dL) in Part A
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part A (Cohort A1, 5 ug Dose) | Part A (Cohort A2, 10 ug Dose) | Part A (Cohort A3, 20 ug Dose) | Part A (Cohort A4, 40 ug Dose) | Part A (Cohort A5, 60 ug Dose) | Part A (Cohort A6, 120 ug Dose) | Part A (Cohort A7, 90 ug Dose) | Part A (Placebo)
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 13
mg/dL | 3.353 (0.6646) | 2.882 (0.3884) | 3.840 (0.5135) | 3.287 (0.5021) | 3.908 (0.5051) | 3.673 (0.4975) | 3.417 (0.4133) | 3.641 (0.3637)

12. Secondary Outcome: Serum Phosphate - Part B
Description: Serum phosphate levels (mg/dL) in Part B
Time Frame: Day 1, Day 14
Population: One (1) subject in Cohort B4 discontinued from the study.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part B (Cohort B1, 10 ug Doses) | Part B (Cohort B2, 20 ug Doses) | Part B (Cohort B3, 40 ug Doses) | Part B (Cohort B4, 60 ug Doses) | Part B (Cohort B5, 80 ug Doses) | Part B (Placebo)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 10
mg/dL
  Day 1 | 3.616 (0.1919) | 3.751 (0.3229) | 3.824 (0.5421) | 3.518 (0.3332) | 3.398 (0.3965) | 3.65 (0.58)
  Day 14: number analyzed (Participants) | 8 | 8 | 8 | 7 | 8 | 10
  Day 14 | 3.601 (0.2299) | 3.850 (0.3397) | 3.603 (0.4738) | 3.727 (0.3970) | 3.553 (0.6037) | 3.74 (0.40)

13. Secondary Outcome: Serum Phosphate - Part C
Description: Serum phosphate levels (mg/dL) in Part C.
Time Frame: Day 1 (H0), Day 14 (H2), Day 28 (H2) and Day 84 (H2)
Population: One (1) subject dropped out in Cohort 2 prior to the extension phase. In addition to this subject, two (2) subjects from Cohort 1 and one (1) subject from Cohort 2 did not participate in the extension phase (data on Day 84). For this reason, data was collected in ten (10) subjects in Cohort 1 and fourteen (14) subjects in Cohort 2 on Day 84. In addition, data not collected for a few subjects (missing data or site error).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part C (Cohort C1, Starting Dose of 20 ug/Day) | Part C (Cohort C2, Starting Dose of 10 ug/Day)
Number analyzed (Participants) | 12 | 16
mg/dL
  Day 1 | 4.12 (0.798) | 4.53 (0.780)
  Day 14: number analyzed (Participants) | 12 | 15
  Day 14 | 3.43 (0.742) | 3.95 (0.849)
  Day 28 | 3.50 (0.843) | 3.82 (0.868)
  Day 84: number analyzed (Participants) | 10 | 14
  Day 84 | 3.60 (0.589) | 3.80 (6.83)

14. Secondary Outcome: Daily Dose of Oral Calcium and Active Vitamin D - Part C
Description: Daily dose of oral calcium and active vitamin D for patients treated in Part C.
Time Frame: Day 28 and Day 43
Population: * One (1) subject dropped out in Cohort 2 prior to the extension phase. In addition to this subject, two (2) subjects from Cohort 1 and one (1) subject from Cohort 2 did not participate in the extension phase (data on Day 84). For this reason, data was collected in ten (10) subjects in Cohort 1 and fourteen (14) subjects in Cohort 2 on Day 84.
  * On Day 84, one (1) patient in Cohort 1 was mistakenly given vitamin D. This patient is included in the nine (9) patients taking no vit D on Day 84.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C (Cohort C1, Starting Dose of 20 ug/Day) | Part C (Cohort C2, Starting Dose of 10 ug/Day)
Number analyzed (Participants) | 12 | 16
Participants
  Number of patients taking =< 500 mg/day of calcium on Day 28 | 9 | 12
  Number of patients taking =< 500 mg/day of calcium on Day 84: number analyzed (Participants) | 10 | 14
  Number of patients taking =< 500 mg/day of calcium on Day 84 | 8 | 13
  Number of patients taking no vitamin D on Day 28 | 10 | 12
  Number of patients taking no vitamin D on Day 84: number analyzed (Participants) | 10 | 14
  Number of patients taking no vitamin D on Day 84 | 9 | 13

15. Other Pre Specified Outcome: Calcium Excretion Rate 24h- Part C
Description: 24 hour calcium excretion rate (mg/24h) in Part C.
Time Frame: Day 1, Day 14, Day 28 and Day 84
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mg/24h
Arm/Group | Part C (Cohort C1, Starting Dose of 20 ug/Day) | Part C (Cohort C2, Starting Dose of 10 ug/Day)
Number analyzed (Participants) | 12 | 16
mg/24h
  Day 1 | 328.72 (130.950) | 330.73 (189.154)
  Day 14 | 224.83 (108.570) | 188.41 (100.054)
  Day 28 | 155.06 (61.705) | 166.43 (96.637)
  Day 84: number analyzed (Participants) | 10 | 14
  Day 84 | 115.70 (37.929) | 145.15 (113.563)

ADVERSE EVENTS:
Time Frame: Up to 2 weeks (Part A and Part B) and up to 3 months (Part C)
Arm/Group | Part A (Cohort A1, 5 ug Dose) | Part A (Cohort A2, 10 ug Dose) | Part A (Cohort A3, 20 ug Dose) | Part A (Cohort A4, 40 ug Dose) | Part A (Cohort A5, 60 ug Dose) | Part A (Cohort A6, 120 ug Dose) | Part A (Cohort A7, 90 ug Dose) | Part A (Placebo) | Part B (Cohort B1, 10 ug Doses) | Part B (Cohort B2, 20 ug Doses) | Part B (Cohort B3, 40 ug Doses) | Part B (Cohort B4, 60 ug Doses) | Part B (Cohort B5, 80 ug Doses) | Part B (Placebo) | Part C (Cohort C1, Starting Dose of 20 ug/Day) | Part C (Cohort C2, Starting Dose of 10 ug/Day)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/13 | 0/8 | 0/8 | 0/10 | 0/8 | 0/8 | 0/10 | 0/12 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/13 | 0/8 | 0/8 | 0/10 | 0/8 | 0/8 | 0/10 | 0/12 | 0/16
Other Adverse Events (participants affected / at risk) | 2/3 | 3/6 | 5/6 | 1/6 | 3/6 | 6/6 | 6/6 | 8/13 | 6/8 | 7/8 | 10/10 | 8/8 | 7/8 | 9/10 | 7/12 | 12/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A (Cohort A1, 5 ug Dose) (N=3) | Part A (Cohort A2, 10 ug Dose) (N=6) | Part A (Cohort A3, 20 ug Dose) (N=6) | Part A (Cohort A4, 40 ug Dose) (N=6) | Part A (Cohort A5, 60 ug Dose) (N=6) | Part A (Cohort A6, 120 ug Dose) (N=6) | Part A (Cohort A7, 90 ug Dose) (N=6) | Part A (Placebo) (N=13) | Part B (Cohort B1, 10 ug Doses) (N=8) | Part B (Cohort B2, 20 ug Doses) (N=8) | Part B (Cohort B3, 40 ug Doses) (N=10) | Part B (Cohort B4, 60 ug Doses) (N=8) | Part B (Cohort B5, 80 ug Doses) (N=8) | Part B (Placebo) (N=10) | Part C (Cohort C1, Starting Dose of 20 ug/Day) (N=12) | Part C (Cohort C2, Starting Dose of 10 ug/Day) (N=16)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Motion Sickness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Otorrhea (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Asthenophenia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bowel Movement Irregularity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Sounds Abdominal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 5 (11) | 4 (5) | 3 (3) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Administration site hematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
application site pruritis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site hematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Catheter site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter Site Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Catheter Site Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hunger (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection Site Bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Injection Site Erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 4 (7) | 3 (7) | 2 (5) | 1 (2) | 1 (1) | 5 (7)
Injection Site Hematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (5) | 5 (11) | 3 (5) | 3 (7) | 3 (4) | 1 (1) | 2 (2)
Injection Site Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Injection Site Pruritis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Injection Site Reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Injection Site Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Puncture site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Odema Peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site hematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Vessel puncture site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asymptomatic COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urine calcium/creatine ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin D increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (7)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 4 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 2 (2)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 4 (6)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 4 (12) | 1 (1) | 3 (5) | 2 (3) | 4 (5)
Hypoasthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (8) | 3 (11) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalciuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sensitive Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT05239221/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-26): https://cdn.clinicaltrials.gov/large-docs/21/NCT05239221/SAP_001.pdf